CLINICAL TRIAL: NCT04108325
Title: A Single-Arm, Open-Label, Multi-Center, Phase Ib Study of YY-20394 in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: A Phase Ib Study of YY-20394 in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-004
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Relapsed or Refractory Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): YY-20394 tablets will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — Each treatment cycle is comprised of 28-day consecutive of YY-20394, 80mg QD (days 1 to 28). Upon completion of each cycle, patients may continue to receive oral YY-20394 tablets if there are benefit from the treatment and the toxicity is tolerable.

SUMMARY:
A single-arm, open, multicenter study to investigate the efficacy and safety of YY-20394, an oral small molecular inhibitor of PI3K-delta, in patients with relapsed or refractory peripheral T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically or cytologically confirmed diagnosis of relapsed or refractory peripheral T cell lymphoma.
3. Eastern Cooperative Oncology Group performance status of 0 to 2.
4. Life expectancy of at least 3 months.
5. At least one measurable lesion according to IRWG.
6. Adequate organ function.
7. Had anti-tumor treatments greater than or equal to 2 weeks prior to the first dose of investigational product (including TKI, chemotherapy, radiotherapy, immunotherapy and major surgery).
8. Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose.
9. Volunteers did not participate in other clinical trials within 1 month prior to study entry.
10. Able to comply with the protocol judged by investigator.
11. Provision of signed and dated, written informed consent prior to any study- specific evaluation.

Exclusion Criteria:

1. Previous treatment with any PI3K-delta ihinibitors. 2. Uncontrolled pleural effusion and ascites. 3. the dosage of steroid hormone ( prednisone equivalent ) was greater than 20mg/day, and lasted for more than 14 days. 4. Medical conditions in swallowing, malabsorption, or other chronic gastrointestinal disease that may hamper compliance and/or absorption of the investigational agent. 5. During the study period, drugs that may prolong the QT (such as anti arrhythmic drugs) could not be interrupted. 6. Evidence of central nervous system involvement of the malignancy, including invasion of brain parenchyma and meninges, or spinal cord compression. 7. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy(such as pneumonia). 8. Active infection with hepatitis B and C virus ( Volunteers with HBsAg or HBcAb positive and HBV-DNA greater than or equal to 1000 coRpies/ml or 200IU/ml; HCV antibody and HCV-RNA positive ). 9. History of immune deficiency ( acquired or congenital ), or history of organ transplantation, or allogeneic bone marrow or hematopoietic stem cell transplantation. 10. Presence of severe or uncontrolled cardiovascular disease. 11. The baseline pregnancy test was positive in pregnant women, lactating women or fertile women. 12. According to the judgement of the investigator, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study (such as severe hypertension, diabetes, thyroid diseases, etc.). 13. Medical history of other primary malignant tumors in the past 5 years except for the following: clinically cured cervical in situ, local basal cell carcinoma of the skin.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 12 months
  Objective Response Rate
DCR | up to 12 months
  Disease control rate
Safety and Tolerability | up to 12 months
  safety and tolerability of investigational product assessed as the number of participants experiencing adverse events (AEs, CTCAE5.0) or abnormalities in vital signs, laboratory tests, or electrocardiograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No